CLINICAL TRIAL: NCT06513975
Title: Validation Study of CART BP as a Wearable Cuffless Blood Pressure Monitor: Evaluation of Blood Pressure Measurement by Height and Physical Activity
Brief Title: Validation Study of CART BP as a Wearable Cuffless Blood Pressure Monitor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sky Labs (Industry)
Collaborators: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SL_BP_V1.0
Record Dates: First submitted 2024-07-16; First posted 2024-07-23 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Blood Pressure; Hypertension; Blood Pressure, High; Blood Pressure, Low; Hypotension
MeSH Terms: conditions — Hypertension; Hypotension | interventions — Sphygmomanometers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects requiring 24-hour ambulatory blood pressure monitoring (Experimental): Subjects prescribed for ambulatory blood pressure monitor (ABPM) measure 24-hour blood pressure using both the CART BP and sphygmomanometer
  Interventions: Device: CART BP; Device: sphygmomanometer

INTERVENTIONS:
Device: CART BP — A ring-type medical device worn by the subject that non-invasively measures systolic and diastolic blood pressure, as well as pulse rate.
Device: sphygmomanometer — Blood pressure measurement method utilizing a two-headed stethoscope, allowing two observers to simultaneously hear the Korotkoff sounds.

SUMMARY:
This study aims to evaluate the accuracy of the CART BP, a medically approved ring-type blood pressure monitor, in comparison to the traditional auscultatory method using a dual-head stethoscope. The comparison is conducted in accordance with the 2023 European Society of Hypertension (ESH) Recommendations, focusing on patients with suspected hypertension or hypotension. The evaluation includes accuracy measurements across various postures and during different exercise periods.

DETAILED DESCRIPTION:
There is a non-invasive technique called Photoplethysmography (PPG) that overcomes the limitations of traditional auscultatory and oscillometric methods. Photoplethysmography uses light-emitting diodes (LEDs) to illuminate human tissue, specifically targeting blood vessels, and employs sensors to measure the volume of blood flowing through the tissue. This technique can be applied to various parts of the small arterial system in the human body, enabling cuffless blood pressure measurement. As a result, it simplifies blood pressure monitoring for subjects and allows for extended observation periods.

With the advancement of cuffless blood pressure monitors, the European Society of Hypertension (ESH) has established recommendations to ensure accurate measurements. The recommendations consider variations in measurement height and compare accuracy after blood pressure is elevated through aerobic exercise or low-intensity repetitive exercises, such as handgrip exercises. This study aims to follow the 2023 European Society of Hypertension recommendations by measuring blood pressure with the arm positioned vertically more than 20 centimeters below the standard position and comparing the results obtained after repeated handgrip exercises with those obtained using the standard method.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 years or older but younger than 80 years
* Individuals who voluntarily decide to participate in this clinical trial and provide written consent to the information and consent form
* Individuals willing to comply with the clinical trial protocol

Exclusion Criteria:

* Subjects who do not consent to the study
* Obese individuals with a Body Mass Index (BMI) of 30 or higher (concerns about measurement errors as the standard 24-hour ambulatory blood pressure monitor cuff may not fit the arm properly)
* Patients or volunteers who are pregnant
* Patients or volunteers with underlying heart diseases: those with a history of hospitalization for heart failure, valvular disease, or myocardial infarction
* Patients or volunteers diagnosed with atrial fibrillation on a 12-lead electrocardiogram (ECG) within the past 6 months
* Patients or volunteers with end-stage renal disease (undergoing dialysis)
* Patients or volunteers unable to perform repeated exercises required for the study
* Patients or volunteers with a systolic blood pressure (SBP) exceeding 160 millimeters of mercury (mmHg)
* Patients or volunteers with a systolic blood pressure (SBP) exceeding 160 millimeters of mercury (mmHg) and/or a diastolic blood pressure (DBP) exceeding 100 millimeters of mercury (mmHg) (for exercise tests)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Mean error and standard deviations of differences between CART BP and Reference | 1 hour
  The primary outcome measure is the mean error and standard deviation (SD) of the differences between the CART BP device and the reference device. This endpoint is determined based on the European Hypertension Society (ESH) recommendation, which states that the pass criteria are as per International Organization for Standardization (ISO) 81060-2:2018: a mean error within 5 mmHg and an standard deviation within ±8 mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Seung Woo Park, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carey RM, Muntner P, Bosworth HB, Whelton PK. Prevention and Control of Hypertension: JACC Health Promotion Series. J Am Coll Cardiol. 2018 Sep 11;72(11):1278-1293. doi: 10.1016/j.jacc.2018.07.008. PMID 30190007
- [Background] Stergiou GS, Avolio AP, Palatini P, Kyriakoulis KG, Schutte AE, Mieke S, Kollias A, Parati G, Asmar R, Pantazis N, Stamoulopoulos A, Asayama K, Castiglioni P, De La Sierra A, Hahn JO, Kario K, McManus RJ, Myers M, Ohkubo T, Shroff SG, Tan I, Wang J, Zhang Y, Kreutz R, O'Brien E, Mukkamala R. European Society of Hypertension recommendations for the validation of cuffless blood pressure measuring devices: European Society of Hypertension Working Group on Blood Pressure Monitoring and Cardiovascular Variability. J Hypertens. 2023 Dec 1;41(12):2074-2087. doi: 10.1097/HJH.0000000000003483. Epub 2023 Jun 22. PMID 37303198
- [Background] Kario K, Shin J, Chen CH, Buranakitjaroen P, Chia YC, Divinagracia R, Nailes J, Hoshide S, Siddique S, Sison J, Soenarta AA, Sogunuru GP, Tay JC, Teo BW, Turana Y, Zhang Y, Park S, Van Minh H, Wang JG. Expert panel consensus recommendations for ambulatory blood pressure monitoring in Asia: The HOPE Asia Network. J Clin Hypertens (Greenwich). 2019 Sep;21(9):1250-1283. doi: 10.1111/jch.13652. PMID 31532913
- [Background] O'Brien E, Parati G, Stergiou G, Asmar R, Beilin L, Bilo G, Clement D, de la Sierra A, de Leeuw P, Dolan E, Fagard R, Graves J, Head GA, Imai Y, Kario K, Lurbe E, Mallion JM, Mancia G, Mengden T, Myers M, Ogedegbe G, Ohkubo T, Omboni S, Palatini P, Redon J, Ruilope LM, Shennan A, Staessen JA, vanMontfrans G, Verdecchia P, Waeber B, Wang J, Zanchetti A, Zhang Y; European Society of Hypertension Working Group on Blood Pressure Monitoring. European Society of Hypertension position paper on ambulatory blood pressure monitoring. J Hypertens. 2013 Sep;31(9):1731-68. doi: 10.1097/HJH.0b013e328363e964. PMID 24029863